CLINICAL TRIAL: NCT03985748
Title: Evaluating the Utilization and Effectiveness of Breath-actuated Nebulizers in Acute COPD Exacerbations
Brief Title: Breath-actuated Nebulizers in Acute COPD Exacerbations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rhode Island Hospital (Other)
Collaborators: Monaghan Medical Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1204420-9
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: COPD Exacerbation
Keywords: Nebulizer; Breath Actuated Nebulizer

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized to receive AeroEclipse® II BAN or SN in the Rhode Island Hospital (RIH) Emergency Department. They will have an equal chance of being placed in either group. Patients will be screened and identified in the Emergency Department. They will receive the BAN or SN for the duration of their stay in the hospital, as long as clinically indicated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Breath Actuated Nebulizers (BAN) (Experimental): Enrolled patients will be randomized to receive AeroEclipse® II BAN or SN in the RIH Emergency Department. They will have an equal chance of being placed in either group. Patients will be screened and identified in the Emergency Department. They will receive the BAN or SN for the duration of their stay in the hospital, as long as clinically indicated.
  Interventions: Device: BAN
- Standard Nebulizer (SN) (Active Comparator): Enrolled patients will be randomized to receive AeroEclipse® II BAN or SN in the RIH Emergency Department. They will have an equal chance of being placed in either group. Patients will be screened and identified in the Emergency Department. They will receive the BAN or SN for the duration of their stay in the hospital, as long as clinically indicated.
  Interventions: Device: SN

INTERVENTIONS:
Device: BAN — Inhaled bronchodilators will be delivered using an AeroEclipse® II Breath Actuated Nebuliz (BAN)
  Arms: Breath Actuated Nebulizers (BAN)
Device: SN — Inhaled bronchodilators will be delivered using a Standard Nebulizer (SN)
  Arms: Standard Nebulizer (SN)

SUMMARY:
The goal of this study is to evaluate the utilization and outcomes of AeroEclipse® II Breath Actuated Nebulizer (BAN, Monaghan Medical Corporation, Plattsburgh, NY) vs. standard continuous flow nebulizers (SN). We hypothesize that the use of AeroEclipse® II BAN will reduce the number of nebulizer treatments needed (primary outcome).

DETAILED DESCRIPTION:
Overview:

Effective administration of aerosolized medications depends on the patient's age, physical and cognitive ability the delivery system, and the patient-device interface. Physical ability means the patient's ability to use a specific device, based on factors such as inspiratory volumes and flows, hand-breath coordination, or ability to use a mouthpiece. Cognitive ability indicates the patient's understanding of how and when to use a device and medication. Airway size, respiratory rate, inspiratory flow rate, and breathing pattern create substantial challenges for effective aerosol delivery. While most aerosol generators can be used with all age groups, special consideration should be given to young children because they cannot master the complex steps required for adequate delivery of aerosol treatments. A mouthpiece may be used for patients > 3 years who are able to cooperate, while a face mask is recommended for patients who cannot use a mouthpiece. Face masks should be properly fitted with minimal leak, particularly avoiding aerosol delivery into the eyes, to optimize inhaled dose. Aerosol generators are equally efficacious if they are age appropriate and used correctly. Regardless of age, patients need to demonstrate ability to seal the lips around the mouthpiece and ability to generate sufficient flow for the specific inhaler. However, the impact of breath-actuation on nebulizer utilization and outcomes vs. standard nebulizer has yet to be evaluated.

Per the American Association Respiratory Care (AARC) Clinical Practice Guidelines for Aerosol Delivery Device Selection for Spontaneously Breathing Patients: 2012, the "appropriate selection of an aerosol generator" is reflected by 1) a positive clinical outcome after aerosol therapy, 2) use of proper technique in applying aerosol delivery system, 3) patient adherence with application of aerosol delivery systems.

Admissions to Rhode Island Hospital (RIH) for respiratory failure due to chronic obstructive pulmonary disease (COPD) exacerbations are common. COPD exacerbations are typically treated with a combination of intravenous or oral corticosteroids and inhaled bronchodilators. Inhaled bronchodilators, including Albuterol, Atrovent and Combivent (a combination of Albuterol and Atrovent), are usually administered as a nebulized solution until there is clinical improvement to the point where patients can be transitioned back to their outpatient metered dose inhalers (MDIs). Standard nebulizers are delivered as a continuous stream of inhaled medication through an interface that the patient holds in his/her mouth. As the medication is delivered irrespective of whether the patient is inhaling or exhaling, a significant portion that is intended to be deposited into the lung never reaches its destination.

Recently, Breath Actuated Nebulizers (BANs) have been developed to provide nebulized medications only when the patient inhales. Industry-sponsored studies, included those that have been funded by Monaghan Medical (Monaghan Medical Corporation, Plattsburgh, NY), the manufacturer of the AeroEclipse II BAN, have demonstrated that nebulized medications delivered via a BAN device have improved drug deposition to more distal areas of the lungs. Patients admitted to the hospital with an acute COPD exacerbation have improved lung hyperinflation and tachypnea when nebulized bronchodilators are administered through a BAN device compared with a continuous flow nebulizer. In addition, BAN use has been associated with a cost savings, in part due to improved workflow efficiency for respiratory therapists and a decrease in the overall number of nebulizer treatments needed. However, there is a paucity of data that address more clinically-relevant outcomes in patients hospitalized with COPD exacerbations that are treated with bronchodilators delivered by BANs versus continuous flow nebulizers.

Specific Aims:

To evaluate the utilization and outcomes of AeroEclipse® II Breath Actuated Nebulizer (BAN, Monaghan Medical Corporation, Plattsburgh, NY) vs. standard continuous flow nebulizers (SN). We hypothesize that the use of AeroEclipse® II BAN will reduce the number of nebulizer treatments needed (primary outcome). Other clinical outcomes gathered (secondary outcomes) are described in Experimental Design and Methods.

Experimental Design and Methods:

This is a prospective, single-center superiority randomized controlled trial. All patients admitted to RIH from the Emergency Department for acute COPD exacerbation are eligible for enrollment. The risks of involvement are no greater than if the patient was not to participate as these patients all receive nebulizers as standard of care. Clinically, either BAN or SN can be utilized in acute COPD exacerbations to delivery aerosolized drugs. Both BAN and SN are FDA approved and are currently marketed. BAN's breath-actuating technology offers more targeted, on-demand drug delivery, which consequently increases the cost of the device. RIH does not currently use the BAN in adult patient care services because the of the lack of available clinical superiority data (the data we are seeking to gather from the present, proposed investigation) to justify such additional costs. The breath-actuating technology uses a one-way valve to deliver the aerosol in response to the patient's inspiratory flow. The SN does not have such a one-way valve, thus delivers the drug in a more continuous, uninterrupted flow.

Enrolled patients will be randomized to receive AeroEclipse® II BAN or SN in the RIH Emergency Department. They will have an equal chance of being placed in either group. Patients will be screened and identified in the Emergency Department. They will receive the BAN or SN for the duration of their stay in the hospital, as long as clinically indicated.

We propose to enroll up to 150 patients to participate in the study for the duration of their stay in the hospital. Consent will be obtained ideally from patients in the Emergency Department although if still eligible, patients could be consented on the patient care unit. The collected data will be obtained specifically for research purposes.

On subject enrollment, the St. George's Respiratory Questionnaire for COPD patients (SGRQ-C) will be administered. The SGRQ is a 14-item questionnaire developed to measure health status (quality of life) in patients with COPD and is well-validated in this patient population. The SGRQ-C will serve as a baseline measurement for each patient. Not all patients at the time of inclusion will have any objective data to support the diagnosis of COPD (i.e., no previous PFTs). Therefore, this information will provide some measurement of disease severity for these patients. Patients will use either BAN or SN per randomization assignment for as long as treatment with nebulizers is clinically indicated by their healthcare team for the duration of their stay in the hospital. If patients get intubated, they will remain enrolled in the study as long as treatment with nebulizers is clinically indicated by their healthcare team after extubation. Researchers will review the patient's EMR for demographic, past medical history, medications, vital signs, nursing data, radiographic, and laboratory data.

Subjects in both groups will have bedside, handheld PFTs performed (measuring FEV1 and FVC) at baseline. These measurements will be performed by respiratory therapist or trained research personnel. Subjects will also be asked to complete a daily Likert scale rating their shortness of breath while receiving nebulizer treatments for up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older and must be admitted to RIH for acute COPD exacerbation
* Patient must be able to understand the information about the research protocol that is provided by the investigators and be able to sign the informed consent form.

  * If a patient does not meet this criterion, consent can be obtained from a surrogate decision maker
  * Spanish speaking patients will be included and consent will be obtained using the short form and an interpreter. The SGRQ-C is translated and validated in Spanish and is readily available.

Exclusion Criteria:

* Patients who are unable or unwilling to receive nebulizer treatments per assigned randomization group
* Inability to enroll patient within 24 hours of presentation to the Emergency Department, where Time 0 = triage time, or before administration of the 5th nebulizer treatment, whichever comes first
* Pregnant women
* Prisoners
* Anyone who uses a BAN as an outpatient
* Patients on continuous BiPAP

  *** These patients usually get nebs administered via an in-line nebulizer device that goes directly into the BiPAP tubing. For those receiving continuous BiPAP, the hand-held BAN cannot be used, as it does not offer an in-line option. In contrast, for those on intermittent BiPAP, patients usually receive hand-held nebulizer, thus remain eligible for BAN, as long as they have the capacity to use the hand-held nebulizer
* Patients who are intubated (orotracheal or nasotracheal) or have a tracheostomy tube *** The hand-held BAN cannot be used for the same reason as for patients on BiPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Total number of nebulizer treatments administered | Through study completion, an average of 6 months
  Medication administration data gathered from electronic medical record (EMR) after patient discharge
Time to nebulizer treatment de-escalation (i.e. standing order to prn order to discontinuation) | Through study completion, an average of 6 months
  Medication administration data gathered from EMR after patient discharge to determine when standing nebulizer orders are changed to as needed (prn) nebulizer orders
Time to return to baseline supplemental oxygen requirement | Through study completion, an average of 6 months
  Supplemental oxygen data gathered from respiratory/nursing flow sheets. For patients not on supplemental oxygen at baseline, time to return to room air

SECONDARY OUTCOMES:
Hospital length of stay (LOS) | Through study completion, an average of 6 months
  Gathered from the EMR hospital course
Need for transfer to a higher level of care and LOS on those units | Through study completion, an average of 6 months
  Gathered from EMR
Progression to intubation/mechanical ventilation | Through study completion, an average of 6 months
  Gathered from EMR
Time requiring non-invasive positive pressure ventilation | Through study completion, an average of 6 months
  Device duration data gathered from EMR Respiratory complications
Discharge location | Through study completion, an average of 6 months
  Where the patient was discharged to after hospitalization (i.e. home, skilled nursing facility, inpatient rehab)
Hospital Mortality | Through study completion, an average of 6 months
  EMR death record
6-month post-discharge data | Through study completion, an average of 6 months
  Access medical records of those that are enrolled for up to 6 months post discharge. This will allow us to obtain PFT reports for patients that did not have PFTs pre-hospitalization and to determine many times subjects are re admitted in 6 months (another secondary outcome)
30-day (+ 7 days) readmission rate | Through study completion, an average of 6 months
  EMR review and/or patient phone contact
Patient-reported ease of device use (USE Questionnaire) | Through study completion, an average of 6 months
  5-10 minutes to complete, completed on study Day 3 (± 1 day)

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03985748/ICF_000.pdf